CLINICAL TRIAL: NCT01696994
Title: Prostate, Lung, Colorectal, and Ovarian (PLCO) Cancer Screening Trial
Brief Title: Screening for Ovarian Cancer in Older Patients (PLCO Screening Trial)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: NCI-2012-01758; NCI-2012-01758 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000078532; NCI-P93-0050; PLCO-1; PLCO-Ovarian (Other: National Cancer Institute)
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Carcinoma; Ovarian Germ Cell Tumor
MeSH Terms: conditions — Ovarian Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Control (No Intervention): Participants receive standard medical care. Participants complete a DHQ at baseline.
- Ovarian Screening (Active Comparator): Participants undergo blood sample collection for CA125 analysis at baseline annually for 5 years. Serum that is not used in the study will be stored in an NCI biorepository. Participants also undergo an OVR (discontinued in December 1998) and TVU at baseline and annually for 3 years. Participants complete a DQX at baseline and DHQ at year 3. An ADU (previously referred to as the PSH questionnaire) is mailed to each participant annually for 13 years to identify all prevalent and incident cancers of the ovaries as all deaths that occur among both screened and control subjects during the trial.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Screening Questionnaire Administration; Procedure: Ultrasound Imaging

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
  Arms: Ovarian Screening
Other: Screening Questionnaire Administration — Undergo questionnaire assessments
  Arms: Ovarian Screening
Procedure: Ultrasound Imaging — Undergo TVU
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US
  Arms: Ovarian Screening

SUMMARY:
This clinical trial studies whether screening methods used to diagnose cancer of the prostate, lung, colon, rectum, or ovaries can reduce deaths from these cancers. Screening tests may help doctors find cancer cells early and plan better treatment for ovarian cancer. The ovarian cancer screening tests are part of a trial that addresses the screening of four cancer sites, each with their own results record: prostate (NCT00002540), lung (NCT01696968), colorectal (NCT01696981), and ovarian (NCT01696994).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether screening with CA125 and transvaginal ultrasound (TVU) can reduce mortality from ovarian cancer in women aged 55-74 at entry.

SECONDARY OBJECTIVES:

I. To assess screening variables, other than mortality, for each of the interventions including sensitivity, specificity, and positive predictive value.

II. To assess the incidence, stage, and survival of cancer cases. III. To investigate the mortality predictive value of biologic and/or prognostic characterizations of tumor tissue as intermediate endpoints.

IV. To conduct biomolecular and genetic research into factors associated with cancer carcinogenesis and promotion, as well as the early detection of these factors.

OUTLINE: Participants in the overall PLCO study are stratified by screening center, gender, and age (55-59 vs 60-64 vs 65-69 vs 70-74). Participants are randomized to 1 of 2 arms (control vs screening).

ARM I (Control): Participants receive standard medical care. Participants complete a Diet History Questionnaire (DHQ) at baseline.

ARM II (Ovarian Screening): Participants undergo blood sample collection for CA125 analysis at baseline annually for 5 years. Serum that is not used in the study will be stored in an NCI biorepository. Participants also undergo an ovarian palpation exam (OVR, discontinued in December 1998) and TVU at baseline and annually for 3 years. A scheduling and tracking procedure is implemented to ensure regular attendance at repeat screens for participants screened negative or for those who are designated suspicious or positive at screening but for whom subsequent diagnostic procedures do not reveal ovarian cancer (follow-up diagnostic procedures are through their own medical care environment). Participants diagnosed with ovarian cancer via a screening test are referred for treatment in accordance with current accepted practice for appropriate stage of disease, patient age, and medical condition; a procedure is provided for contact with qualified medical personnel to insure appropriate therapy.

Participants complete a Dietary Questionnaire (DQX) at baseline and DHQ at year 3. An Annual Study Update (ADU) (previously referred to as the Periodic Survey of Health [PSH] questionnaire) is mailed to each participant annually for 13 years to identify all prevalent and incident cancers of the ovaries as all deaths that occur among both screened and control subjects during the trial.

After completion of screening, participants are followed up for at least 13 years.

ELIGIBILITY:
Exclusion Criteria:

* Women who at the time of randomization are less than 55 or greater than or equal to 75 years of age
* Individuals undergoing treatment for cancer at this time, excluding basal-cell and squamous-cell skin cancer
* Individuals with known prior cancer of the colon, rectum, lung, or ovary

  * This includes primary or metastatic PLCO cancers
* Individuals with previous surgical removal of the entire colon or one lung

  * Until October 1996, women with previous surgical removal of both ovaries were excluded from the trial. In order to increase the enrollment of women into the trial, beginning in October 1996, these women were no longer excluded for this reason.
* Individuals who are participating in another cancer screening or cancer primary prevention trial
* Prior to April 1, 1999 women were excluded from the trial if they were currently taking or had taken Tamoxifen or Evista\Raloxifene in the past 6 months. As of April 1999 based on a decision from the PLCO Ovary Subcommittee, women who have or are currently taking Tamoxifen or Evista\Raloxifene are not excluded from participation.
* Individuals who are unwilling or unable to sign the informed consent form
* Individuals who have had a colonoscopy, sigmoidoscopy, or barium enema in the past three years

Ages: 55 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78216 (Actual)
Dates: Start 1993-11-16 (Actual); Primary Completion 2012-05-21 (Actual); Study Completion 2026-03-25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christine D Berg, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Malcomson FC, Shams-White MM, Reedy J, Huang WY, Moore SC, Loftfield E. Adherence to the 2018 World Cancer Research Fund/American Institute for Cancer Research Cancer Prevention Recommendations and risk of lifestyle-related cancers in the prostate, lung, colorectal, and ovarian cancer screening trial. BJC Rep. 2025 Nov 19;3(1):81. doi: 10.1038/s44276-025-00195-6. PMID 41261199
- [Derived] Fan Z, Zhang Y, Yao Q, Liu X, Duan H, Liu Y, Sheng C, Lyu Z, Yang L, Song F, Huang Y, Song F. Effects of joint screening for prostate, lung, colorectal, and ovarian cancer - results from a controlled trial. Front Oncol. 2024 Apr 29;14:1322044. doi: 10.3389/fonc.2024.1322044. eCollection 2024. PMID 38741776
- [Derived] Jiang Y, Xie Q, Chen R. Breast Cancer Incidence and Mortality in Relation to Hormone Replacement Therapy Use Among Postmenopausal Women: Results From a Prospective Cohort Study. Clin Breast Cancer. 2022 Feb;22(2):e206-e213. doi: 10.1016/j.clbc.2021.06.010. Epub 2021 Jun 26. PMID 34548240
- [Derived] Wang K, Wu Q, Li Z, Reger MK, Xiong Y, Zhong G, Li Q, Zhang X, Li H, Foukakis T, Xiang T, Zhang J, Ren G. Vitamin K intake and breast cancer incidence and death: results from a prospective cohort study. Clin Nutr. 2021 May;40(5):3370-3378. doi: 10.1016/j.clnu.2020.11.009. Epub 2020 Nov 16. PMID 33277073

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between November 1993 and July 2001 at 10 study centers.
Pre-assignment Details: Participants signed a study informed consent prior to being randomized to a study arm.
Groups:
- Control: Participants receive standard medical care.
- Ovarian Screening: Participants undergo blood sample collection for CA-125 analysis at baseline annually for 5 years. Participants also undergo an OVR (discontinued in December 1998) and TVU at baseline and annually for 3 years.
Period: Overall Study
Arm/Group | Control | Ovarian Screening
Started | 39111 | 39105
Completed | 33919 | 30668
Not Completed | 5192 | 8437
Not completed — Cancer Before Rand. (Ovarian Screening) | 0 | 2
Not completed — Died Before Randomization | 1 | 2
Not completed — Died Before ASU (Control) | 73 | 0
Not completed — No Ovaries at Baseline | 4807 | 4851
Not completed — Refused ASU (Control) | 311 | 0
Not completed — Refused Screen (Ovarian Screening) | 0 | 3582

BASELINE CHARACTERISTICS:
Groups:
- Control: Participants receive standard medical care. Participants complete a baseline questionnaire (BQ) at entry and a dietary history questionnaire (DHQ) during study years 0-6.
- Ovarian Screening: Participants undergo blood sample collection for Cancer Antigen 125 (CA-125) analysis at baseline and annually for 5 years. Participants also undergo an OVR (discontinued in December 1998) and TVU at baseline and annually for 3 years.
- Total: Total of all reporting groups
Arm/Group | Control | Ovarian Screening | Total
Number analyzed (Participants) | 39111 | 39105 | 78216
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25222 | 25233 | 50455
  >=65 years | 13889 | 13872 | 27761
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (5.4) | 62.5 (5.4) | 62.5 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39111 | 39105 | 78216
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39111 | 39105 | 78216

OUTCOME MEASURES:

1. Primary Outcome: Ovarian Cancer Deaths (Including Primary Peritoneal and Fallopian Tube Cancers)
Description: Ovarian cancer deaths confirmed in participants by a death review committee if available, otherwise by death certificate.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 11.9 years.
Measure: Number; unit: Participants
Arm/Group | Control | Ovarian Screening
Number analyzed (Participants) | 34304 | 34253
Participants | 100 | 188

2. Secondary Outcome: Deaths From All Causes
Description: Deaths from all causes were compared between the ovarian cancer screening arm and the usual care arm.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 11.9 years.
Measure: Number; unit: Participants
Arm/Group | Control | Ovarian Screening
Number analyzed (Participants) | 34304 | 34253
Participants | 3542 | 3508

3. Secondary Outcome: Death Rates From All Causes
Description: Deaths from all causes were compared between the ovarian cancer screening arm and the usual care arm. Rate is the number of deaths divided by person years of follow-up in the study.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 11.9 years.
Population: Female participants, excluding females without ovaries at baseline, were analyzed. An intention-to-treat analysis was performed.
Measure: Number; unit: Deaths per 10,000 PY
Groups:
- Ovarian Screening: Participants undergo blood sample collection for CA125 analysis at baseline annually for 5 years. Participants also undergo an OVR (discontinued in December 1998) and TVU at baseline and annually for 3 years.
Arm/Group | Control | Ovarian Screening
Number analyzed (Participants) | 34304 | 34253
Deaths per 10,000 PY | 92.6 | 91.9
Statistical Analysis 1: Comparison: Control; Test type: Superiority or Other; Poisson regression; Two-sided. Not adjusted for multiple comparisons. A-priori threshold for significance 0.05; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.95 to 1.04]

4. Secondary Outcome: Ovarian Cancer Incidence (Including Primary Peritoneal and Fallopian Tube Cancers)
Description: Ovarian cancer diagnoses confirmed by medical record abstraction.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 11.9 years.
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Control | Ovarian Screening
Number analyzed (Participants) | 34304 | 34253
Participants | 176 | 212

5. Secondary Outcome: Ovarian Cancer Incidence Rates (Including Primary Peritoneal and Fallopian Tube Cancers).
Description: Ovarian cancer diagnoses confirmed by medical record abstraction. Incidence rate (cumulative) defined as ovarian cancer diagnoses divided by person years at risk for ovarian cancer.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 11.9 years.
Population: as for outcome 3
Measure: Number; unit: Diagnoses per 10,000 PY
Arm/Group | Control | Ovarian Screening
Number analyzed (Participants) | 34304 | 34253
Diagnoses per 10,000 PY | 4.7 | 5.7
Statistical Analysis 1: Comparison: Control vs Ovarian Screening; Test type: Superiority or Other; Poisson regression; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.99 to 1.48]

6. Secondary Outcome: Complications of Diagnostic Evaluation (DE) Following a Positive Screening Test
Description: Number of positive screens with complications
Time Frame: One year from screening examination
Population: The units analyzed were positive screening exams with documented diagnostic follow-up. If a participant received 3 positive screens with documented follow-up after each one, she would be counted 3 times in the number of units analyzed.
Measure: Number; unit: Positive screens w/ complications
Units Other Than Participants: Positive Screens with Follow-up
Arm/Group | Ovarian Screening
Number analyzed (Participants) | 3531
Number analyzed (Positive Screens with Follow-up) | 5970
Positive screens w/ complications
  When DE Led to Ovarian Cancer Diagnosis | 49
  When DE Did Not Lead to Ovarian Cancer Diagnosis | 226

7. Secondary Outcome: T0 (Baseline) CA-125 Screening Results
Description: Cancer Antigen 125 (CA-125) result.
Time Frame: T0 (at study entry)
Population: Females in the Ovarian Screening arm (excluding females with no ovaries at baseline) who had a CA-125 screen at T0 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ovarian Screening
Number analyzed (Participants) | 28733
Participants
  Negative (<35 U/mL) | 28275
  Positive (>= 35 U/mL) | 400
  Inadequate screen | 58

8. Secondary Outcome: T0 (Baseline) TVU Screening Results
Description: Transvaginal Ultrasound (TVU) result.
Time Frame: T0 (at study entry)
Population: Females in the Ovarian Screening arm (excluding females with no ovaries at baseline) who had a TVU screen at T0 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ovarian Screening
Number analyzed (Participants) | 28477
Participants
  Negative | 26624
  Positive | 1309
  Inadequate screen | 544

9. Secondary Outcome: T1 CA-125 Screening Results
Description: Cancer Antigen 125 (CA-125) result.
Time Frame: T1 (one year after entry)
Population: Females in the Ovarian Screening arm (excluding females with no ovaries at baseline) who had a CA-125 screen at T1 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ovarian Screening
Number analyzed (Participants) | 27514
Participants
  Negative (<35 U/mL) | 27035
  Positive (>= 35 U/mL) | 433
  Inadequate screen | 46

10. Secondary Outcome: T1 TVU Screening Results
Description: Transvaginal Ultrasound (TVU) result.
Time Frame: T1 (one year after entry)
Population: Females in the Ovarian Screening arm (excluding females with no ovaries at baseline) who had a TVU screen at T1 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ovarian Screening
Number analyzed (Participants) | 27046
Participants
  Negative | 25740
  Positive | 930
  Inadequate screen | 376

11. Secondary Outcome: T2 CA-125 Screening Results
Description: Cancer Antigen 125 (CA-125) result.
Time Frame: T2 (two years after entry)
Population: Females in the Ovarian Screening arm (excluding females with no ovaries at baseline) who had a CA-125 screen at T2 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ovarian Screening
Number analyzed (Participants) | 26555
Participants
  Negative (<35 U/mL) | 26024
  Positive (>= 35 U/mL) | 480
  Inadequate screen | 51

12. Secondary Outcome: T2 TVU Screening Results
Description: Transvaginal Ultrasound (TVU) result.
Time Frame: T2 (one year after entry)
Population: Females in the Ovarian Screening arm (excluding females with no ovaries at baseline) who had a TVU screen at T2 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ovarian Screening
Number analyzed (Participants) | 26048
Participants
  Negative | 24988
  Positive | 764
  Inadequate screen | 296

13. Secondary Outcome: T3 CA-125 Screening Results
Description: Cancer Antigen 125 (CA-125) result.
Time Frame: T3 (three years after entry)
Population: Females in the Ovarian Screening arm (excluding females with no ovaries at baseline) who had a CA-125 screen at T3 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ovarian Screening
Number analyzed (Participants) | 25401
Participants
  Negative (<35 U/mL) | 24925
  Positive (>= 35 U/mL) | 427
  Inadequate screen | 49

14. Secondary Outcome: T3 TVU Screening Results
Description: Transvaginal Ultrasound (TVU) result.
Time Frame: T3 (three years after entry)
Population: Females in the Ovarian Screening arm (excluding females with no ovaries at baseline) who had a TVU screen at T3 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ovarian Screening
Number analyzed (Participants) | 24949
Participants
  Negative | 23926
  Positive | 733
  Inadequate screen | 290

15. Primary Outcome: Ovarian Cancer Death Rates (Including Primary Peritoneal and Fallopian Tube Cancers)
Description: Ovarian cancer deaths confirmed in participants by a death review committee if available, otherwise by death certificate. Rate is the number of deaths divided by person years of follow-up in the study.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 11.9 years.
Population: as for outcome 3
Measure: Number; unit: Deaths per 10,000 PY
Arm/Group | Control | Ovarian Screening
Number analyzed (Participants) | 34304 | 34253
Deaths per 10,000 PY | 2.6 | 3.1
Statistical Analysis 1: Comparison: Control vs Ovarian Screening; Test type: Superiority or Other; Poisson regression — Two-sided. Not adjusted for multiple comparisons. A-priori threshold for significance 0.05; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [.91 to 1.54]

16. Secondary Outcome: T4 CA-125 Screening Results
Description: Cancer Antigen 125 (CA-125) result.
Time Frame: T4 (four years after entry)
Population: Females in the Ovarian Screening arm (excluding females with no ovaries at baseline) who had a CA-125 screen at T4 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ovarian Screening
Number analyzed (Participants) | 20115
Participants
  Negative (<35 U/mL) | 19772
  Positive (>= 35 U/mL) | 327
  Inadequate screen | 16

17. Secondary Outcome: T5 CA-125 Screening Results
Description: Cancer Antigen 125 (CA-125) result.
Time Frame: T5 (five years after entry)
Population: Females in the Ovarian Screening arm (excluding females with no ovaries at baseline) who had a CA-125 screen at T5 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ovarian Screening
Number analyzed (Participants) | 22193
Participants
  Negative (<35 U/mL) | 21788
  Positive (>= 35 U/mL) | 366
  Inadequate screen | 39

ADVERSE EVENTS:
Time Frame: During each annual screening visit.
Description: These events are solely those prompted by the screening examination.
Arm/Group | Ovarian Screening
Serious Adverse Events (participants affected / at risk) | 0/34253
Other Adverse Events (participants affected / at risk) | 903/34253
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ovarian Screening (N=34253)
Anxiety (General disorders) | 3 (3)
Bleeding (General disorders) | 26 (27)
Dizzy (General disorders) | 80 (82)
Fainted (General disorders) | 29 (31)
Inflammation (General disorders) | 2 (2)
Nausea (General disorders) | 4 (4)
Pain (General disorders) | 26 (26)
Bruising (General disorders) | 446 (453)
Hematoma (General disorders) | 284 (292)
Other Adverse Event (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less